CLINICAL TRIAL: NCT03625323
Title: TACTI-002 (Two ACTive Immunotherapeutics): A Multicenter, Open Label, Phase II Study in Patients With Previously Untreated Unresectable or Metastatic Non-small Cell Lung Cancer (NSCLC), or Recurrent PD-X Refractory NSCLC or With Recurrent or Metastatic Squamous Head and Neck Cancer (HNSCC) Receiving the Soluble LAG-3 Fusion Protein Eftilagimod Alpha (IMP321) in Combination With Pembrolizumab (PD-1 Antagonist)
Brief Title: Combination Study With Soluble LAG-3 Fusion Protein Eftilagimod Alpha (IMP321) and Pembrolizumab in Patients With Previously Untreated Unresectable or Metastatic NSCLC, or Recurrent PD-X Refractory NSCLC or With Recurrent or Metastatic HNSCC
Acronym: TACTI-002
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Immutep S.A.S. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TACTI-002; Keynote-MK-3475-798 (Other: Merck Sharp & Dohme LLC); 2018-001994-25 (EudraCT Number)
Record Dates: First submitted 2018-07-16; First posted 2018-08-10 (Actual); Results first posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: NSCLC; HNSCC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — soluble LAG-3 protein, human; pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 1st line NSCLC (Experimental): eftilagimod alpha: 30 mg every 2 weeks for the first 8 cycles (1 cycle = 3 weeks) and every 3 weeks thereafter (starting cycle 9).
  pembrolizumab (KEYTRUDA®): 200 mg every 3 weeks.
  Interventions: Drug: eftilagimod alpha; Drug: pembrolizumab (KEYTRUDA®)
- 2nd line NSCLC (Experimental): eftilagimod alpha: 30 mg every 2 weeks for the first 8 cycles (1 cycle = 3 weeks) and every 3 weeks thereafter (starting cycle 9).
  pembrolizumab (KEYTRUDA®): 200 mg every 3 weeks.
  Interventions: Drug: eftilagimod alpha; Drug: pembrolizumab (KEYTRUDA®)
- HNSCC (Experimental): eftilagimod alpha: 30 mg every 2 weeks for the first 8 cycles (1 cycle = 3 weeks) and every 3 weeks thereafter (starting cycle 9).
  pembrolizumab (KEYTRUDA®): 200 mg every 3 weeks.
  Interventions: Drug: eftilagimod alpha; Drug: pembrolizumab (KEYTRUDA®)

INTERVENTIONS:
Drug: eftilagimod alpha — APC activator, MHC II agonist, LAG-3 fusion protein
  Other Names: IMP321; efti; eftilagimod alfa
Drug: pembrolizumab (KEYTRUDA®) — anti-PD-1 antibody
  Other Names: MK-3475

SUMMARY:
Evaluate the safety and efficacy of the combination of eftilagimod alpha with pembrolizumab in non-small cell lung carcinoma and head and neck carcinoma patients.

DETAILED DESCRIPTION:
Up to 187 patients will be recruited in the TACTI-002 (Two ACTive Immunotherapies) Phase II study which will take place across approximately 22 study centres in the U.S., Europe and Australia. It will evaluate the safety and efficacy of the combination of eftilagimod alpha with pembrolizumab in patients with advanced or metastatic non-small cell lung carcinoma or head and neck carcinoma. It will be a Simon's two-stage, non-comparative, open-label, single-arm, multicentre clinical study. Patients participating in the trial will be given the combination treatment for 12 months using a 30 mg s.c. eftilagimod alpha dosing every 2 or 3 weeks.

ELIGIBILITY:
Main Inclusion Criteria:

1. Part A (1st line, PD-X naïve NSCLC): histologically- or cytologically-confirmed diagnosis of non-small cell lung carcinoma stage IIIB not amenable to curative treatment or stage IV not amenable to EGFR/ALK based therapy, treatment naïve for systemic therapy given for advanced/metastatic disease (previous palliative radiotherapy for advanced/metastatic disease acceptable)

   Part B (2nd line, PD-X refractory NSCLC): histologically- or cytologically-confirmed diagnosis of NSCLC after failure of first-line treatment (for metastatic disease) with at least 2 cycles of any PD-1/PD-L1 containing based therapy (e.g. nivolumab, pembrolizumab, avelumab, durvalumab, etc.) alone, or in combination with any other immunotherapeutic or chemotherapy given as part of first-line treatment.

   Part C (2nd line PD-X naive HNSCC): Histologically- or cytologically-confirmed recurrent disease not amenable to curative treatment with local or systemic therapy, or metastatic (disseminated) HNSCC of the oral cavity, oropharynx, hypopharynx, and larynx that is considered incurable by local therapies after failure of prior platinum-based therapy.
2. Submission of formalin-fixed diagnostic tumor tissue
3. ECOG performance status 0-1.
4. Expected survival > 3 months.

Main Exclusion Criteria:

1. For part A (1st line, PD-X naïve NSCLC):

   * The NSCLC can be treated with curative intent with either surgical resection and/or chemoradiation and/or radiation.
   * Has received systemic therapy for the treatment of their stage IV NSCLC. Completion of treatment with chemotherapy and/or radiation as part of neoadjuvant/adjuvant therapy is allowed as long as therapy was completed at least 6 months prior to the diagnosis of metastatic disease.
   * EGFR-sensitizing mutation and/or is EML4 gene/ ALK gene fusion positive (ALK translocation).
   * Lung radiation therapy that is >30Gy within 6 months of the first dose of trial treatment.

   For Part B (2nd line, PD-X refractory NSCLC):
   * Symptomatic ascites or pleural effusion.
   * > 1 line of chemotherapy for metastatic disease.
   * Lung radiation therapy that is >30Gy within 6 months of the first dose of trial treatment.

   For Part C (2nd line PD-X naive HNSCC):
   * Disease is suitable for local therapy administered with curative intent.
   * Previously treated with > 1 systemic regimens for recurrent and/or metastatic disease.
2. Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways) (Part A and C only)
3. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137) and was discontinued from that treatment due to a Grade 3 or higher irAE (Part B only)
4. Has received prior chemotherapy, anti-cancer monoclonal antibody, major surgery, another systemic cancer therapy or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to cycle 1 day 1.

   Note: Patients must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Patients with ≤Grade 2 neuropathy, alopecia and elevated transaminases in case of liver metastases may be eligible. If patient received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment. Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
5. Known active central nervous system metastasis and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are radiologically stable: i.e. without evidence of progression documented by repeat imaging performed after therapy completed for CNS metastasis and with at least 4 weeks difference, clinically stable and without requirement for steroid treatment for at least 14 days prior to cycle 1 day 1.
6. Receives continuous systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 7 days prior to cycle 1 day 1. Inhaled or topical steroids and physiological replacement doses of up to 10 mg daily prednisone equivalents are permitted in the absence of active auto-immune disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2024-11-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Oncology Consultants, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Krebs MG, Forster M, Majem M, Peguero J, Iams W, Clay T, Roxburgh P, Doger B, Bajaj P, Barba A, Perera S, Mueller C, Triebel F. Eftilagimod Alpha (a Soluble LAG-3 Protein) Combined With Pembrolizumab in Second-Line Metastatic NSCLC Refractory to Anti-Programmed Cell Death Protein 1/Programmed Death-Ligand 1-Based Therapy: Final Results from a Phase 2 Study. JTO Clin Res Rep. 2024 Aug 30;5(11):100725. doi: 10.1016/j.jtocrr.2024.100725. eCollection 2024 Nov. PMID 39403626

RESULTS

PARTICIPANT FLOW:
Groups:
- 1st Line NSCLC; 2nd Line NSCLC; 2nd Line HNSCC: Eftilagimod alpha: 30 mg every 2 weeks for the first 8 cycles (1 cycle = 3 weeks) and every 3 weeks thereafter (starting cycle 9).
  Pembrolizumab: 200 mg every 3 weeks.
  Eftilagimod alpha: APC activator, MHC II agonist, LAG-3 fusion protein
  Pembrolizumab: anti-PD-1 antibody
Period: Overall Study
Arm/Group | 1st Line NSCLC | 2nd Line NSCLC | 2nd Line HNSCC
Started | 114 | 36 | 37
Completed | 0 | 0 | 0
Not Completed | 114 | 36 | 37

BASELINE CHARACTERISTICS:
Groups:
- HNSCC: Eftilagimod alpha: 30 mg every 2 weeks for the first 8 cycles (1 cycle = 3 weeks) and every 3 weeks thereafter (starting cycle 9).
  Pembrolizumab: 200 mg every 3 weeks.
  Eftilagimod alpha: APC activator, MHC II agonist, LAG-3 fusion protein
  Pembrolizumab: anti-PD-1 antibody
- Total: Total of all reporting groups
Arm/Group | 1st Line NSCLC | 2nd Line NSCLC | HNSCC | Total
Number analyzed (Participants) | 114 | 36 | 37 | 187
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 39 | 15 | 20 | 74
  >=65 years | 75 | 21 | 17 | 113
Age, Continuous [Median (Full Range); unit: Years] | 67 [44 to 85] | 67 [46 to 84] | 63 [48 to 84] | 67 [44 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 14 | 4 | 48
  Male | 84 | 22 | 33 | 139
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 1 | 10
  Not Hispanic or Latino | 109 | 32 | 36 | 177
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 0 | 4
  White | 109 | 34 | 35 | 178
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 1 | 3
Smoking history [Count of Participants; unit: Participants]
  Non-smoker | 6 | 5 | 5 | 16
  Ex- or current smoker | 108 | 31 | 32 | 171

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Objective Response Rate (ORR) According to iRECIST (Unconfirmed)
Description: ORR was defined as the percentage of participants for each dose level whose best overall response is rated as iCR or iPR per immune Response Evaluation Criteria In Solid Tumors (iRECIST) for target lesions and assessed by CT or MRI.
  iCR was defined as disappearance of all target and non-target lesions and any pathological lymph nodes must be <10 mm in the short axis.
  iPR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters.
Time Frame: Data collected from screening until time of disease progression, death, lost to follow up, study discontinuation, whichever occurs first, assessed up to approximately 68 months
Measure: Count of Participants; unit: Participants
Arm/Group | 1st Line NSCLC | 2nd Line NSCLC | HNSCC
Number analyzed (Participants) | 114 | 36 | 37
Participants | 46 | 3 | 11

2. Primary Outcome: Evaluation of Objective Response Rate (ORR) According to iRECIST (Confirmed)
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 1st Line NSCLC | 2nd Line NSCLC | HNSCC
Number analyzed (Participants) | 114 | 36 | 37
Participants | 40 | 3 | 10

3. Secondary Outcome: Duration of (Serious) Adverse Events
Time Frame: up to 27 months
Reporting Status: Not Posted

4. Secondary Outcome: Frequency of (Serious) Adverse Events
Time Frame: up to 27 months
Reporting Status: Not Posted

5. Secondary Outcome: Severity of (Serious) Adverse Events
Time Frame: up to 27 months
Reporting Status: Not Posted

6. Secondary Outcome: Time to Responses According to iRECIST and RECIST 1.1
Time Frame: up to 68 months
Reporting Status: Not Posted

7. Secondary Outcome: Duration of Responses According to iRECIST and RECIST 1.1
Time Frame: up to 68 months
Reporting Status: Not Posted

8. Secondary Outcome: Response Rate According to RECIST 1.1
Time Frame: up to 68 months
Reporting Status: Not Posted

9. Secondary Outcome: Disease Control Rate According to iRECIST and RECIST 1.1
Time Frame: up to 68 months
Reporting Status: Not Posted

10. Secondary Outcome: Progression Free Survival (PFS)
Time Frame: up to 68 months
Reporting Status: Not Posted

11. Secondary Outcome: Overall Survival (OS)
Time Frame: up to 68 months
Reporting Status: Not Posted

12. Secondary Outcome: Occurrence of Eftilagimod Alpha-specific Antibodies (ADA)
Time Frame: up to 24 month
Reporting Status: Not Posted

13. Secondary Outcome: Plasma Concentration Time Profile of Eftilagimod Alpha
Time Frame: up to 24 month
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 27 months
Arm/Group | 1st Line NSCLC | 2nd Line NSCLC | 2nd Line HNSCC
All-Cause Mortality (participants affected / at risk) | 14/114 | 2/36 | 7/37
Serious Adverse Events (participants affected / at risk) | 50/114 | 7/36 | 20/37
Other Adverse Events (participants affected / at risk) | 114/114 | 35/36 | 36/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1st Line NSCLC (N=114) | 2nd Line NSCLC (N=36) | 2nd Line HNSCC (N=37)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 2 | 0 | 2
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 3 | 0 | 0
Death (unknown cause) (General disorders) | 3 | 0 | 0
COVID-19 (Infections and infestations) | 2 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 2
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Syncope (Nervous system disorders) | 0 | 0 | 2
Anemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Cardiac failure (Cardiac disorders) | 2 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0
Seizure (Nervous system disorders) | 1 | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 1 | 1
Achromobacter infection (Infections and infestations) | 1 | 0 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1
Endocarditis enterococcal (Infections and infestations) | 0 | 0 | 1
Otitis media (Infections and infestations) | 1 | 0 | 0
Pleural infection (Infections and infestations) | 1 | 0 | 0
Pneumonia viral (Infections and infestations) | 1 | 0 | 0
Prostate infection (Infections and infestations) | 0 | 0 | 1
Pulmonary sepsis (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Immune-mediated pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Atrial thrombosis (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
Gait disturbance (General disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0
Arterial thrombosis (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Biopsy lymph gland (Investigations) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1st Line NSCLC (N=114) | 2nd Line NSCLC (N=36) | 2nd Line HNSCC (N=37)
Asthenia (General disorders) | 37 | 8 | 8
Fatigue (General disorders) | 25 | 7 | 6
Pyrexia (General disorders) | 14 | 2 | 2
Oedema peripheral (General disorders) | 11 | 5 | 0
Injection site pain (General disorders) | 10 | 5 | 0
Injection site erythema (General disorders) | 8 | 5 | 0
Non-cardiac chest pain (General disorders) | 8 | 5 | 0
Injection site reaction (General disorders) | 7 | 4 | 0
Injection site swelling (General disorders) | 4 | 3 | 0
Injection site pruritus (General disorders) | 4 | 2 | 0
Chest pain (General disorders) | 1 | 2 | 0
Facial pain (General disorders) | 1 | 0 | 2
Pain (General disorders) | 1 | 0 | 2
Face oedema (General disorders) | 0 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 40 | 11 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 31 | 11 | 7
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 18 | 1 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 9 | 3 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 19 | 5 | 4
Constipation (Gastrointestinal disorders) | 20 | 4 | 2
Diarrhoea (Gastrointestinal disorders) | 18 | 2 | 5
Vomiting (Gastrointestinal disorders) | 12 | 4 | 3
Dysphagia (Gastrointestinal disorders) | 7 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 5 | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 7 | 2 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 1 | 4
Dry mouth (Gastrointestinal disorders) | 6 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 | 6 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 3 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 13 | 4 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 2 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 8 | 1 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 5 | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 28 | 12 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 9 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 2 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 3 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Pneumonia (Infections and infestations) | 10 | 3 | 2
Upper respiratory tract infection (Infections and infestations) | 4 | 3 | 5
Urinary tract infection (Infections and infestations) | 6 | 1 | 3
COVID-19 (Infections and infestations) | 7 | 0 | 1
Bronchitis (Infections and infestations) | 5 | 1 | 2
Oral candidiasis (Infections and infestations) | 4 | 1 | 2
Respiratory tract infection (Infections and infestations) | 3 | 1 | 3
Skin infection (Infections and infestations) | 5 | 0 | 2
Lower respiratory tract infection (Infections and infestations) | 2 | 2 | 1
Rhinitis (Infections and infestations) | 2 | 2 | 0
Weight decreased (Investigations) | 6 | 6 | 7
Amylase increased (Investigations) | 13 | 2 | 1
Aspartate aminotransferase increased (Investigations) | 6 | 2 | 3
Alanine aminotransferase increased (Investigations) | 6 | 2 | 1
Blood creatinine increased (Investigations) | 6 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 25 | 5 | 4
Rash (Skin and subcutaneous tissue disorders) | 17 | 1 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 8 | 1 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Headache (Nervous system disorders) | 7 | 4 | 2
Dizziness (Nervous system disorders) | 7 | 3 | 2
Paraesthesia (Nervous system disorders) | 4 | 2 | 0
Syncope (Nervous system disorders) | 1 | 1 | 3
Anaemia (Blood and lymphatic system disorders) | 25 | 2 | 7
Hypothyroidism (Endocrine disorders) | 10 | 1 | 8
Hyperthyroidism (Endocrine disorders) | 6 | 0 | 0
Insomnia (Psychiatric disorders) | 11 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 7 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 1 | 3
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 0 | 3
Hypotension (Vascular disorders) | 6 | 0 | 4
Hypertension (Vascular disorders) | 4 | 0 | 3
Urinary retention (Renal and urinary disorders) | 0 | 0 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Approval from the Sponsor is required for the PI to publish or disseminate results from the medical investigation.

DOCUMENTS (2):
  • Study Protocol (2023-08-18): https://cdn.clinicaltrials.gov/large-docs/23/NCT03625323/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-31): https://cdn.clinicaltrials.gov/large-docs/23/NCT03625323/SAP_001.pdf